CLINICAL TRIAL: NCT00277914
Title: 12-month Sustained Efficacy of Flibanserin v Placebo n Younger Women With HSDD in NA
Brief Title: Flibanserin Randomized Withdrawal Trial in Pre-menopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sprout Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 511.74
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Sexual Dysfunctions, Psychological
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — flibanserin

INTERVENTIONS:
Drug: Flibanserin — flibanserin flexible dosing

SUMMARY:
To estimate the duration of efficacy with continued treatment of double-blind flibanserin or placebo over twenty-four weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Women over 18 and pre-menopausal
2. FSDS-R above 14
3. Willingness to try to have sexual activity at least monthly
4. Willingness to use an electronic diary daily
5. Stable, monogamous, heterosexual relationship for at least one year
6. Medically acceptable method of contraception

Exclusion Criteria:

1. Clinically relevant conditions which might interfere with the patient's abil ity to participate in the trial
2. Specified medications
3. Sexual function affected by medication
4. Drug dependence or abuse
5. Sexual partner needing treatment
6. Peri-Menopause or Menopause (surgical or otherwise)
7. Pregnancy
8. Pelvic Inflammatory Disease
9. Major depressive Episode
10. Significant ECG abnormalities
11. Significant Neurologic findings
12. Significant GI, Hepatic, Cardiovascular, Renal, Hematologic, Immunologic or Respiratory findings
13. Uncorrected thyroid or endocrine disease
14. Uncontrolled Glaucoma

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 749 (Actual)
Dates: Start 2006-01; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Duration of efficacy of flibanserin in Sexually Satisfying Events | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (65):
- United States (55):
  - 511.74.01051 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 511.74.01027 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 511.74.01029 Boehringer Ingelheim Investigational Site, Scottsdale, Arizona
  - 511.74.01031 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 511.74.01004 Boehringer Ingelheim Investigational Site, Jonesboro, Arkansas
  - 511.74.01053 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 511.74.01033 Boehringer Ingelheim Investigational Site, Palm Springs, California
  - 511.74.01003 Boehringer Ingelheim Investigational Site, Palo Alto, California
  - 511.74.01015 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 511.74.01013 Boehringer Ingelheim Investigational Site, San Diego, California
  - 511.74.01052 Boehringer Ingelheim Investigational Site, Torrance, California
  - 511.74.01022 Boehringer Ingelheim Investigational Site, Aurora, Colorado
  - 511.74.01046 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 511.74.01002 Boehringer Ingelheim Investigational Site, Groton, Connecticut
  - 511.74.01023 Boehringer Ingelheim Investigational Site, Middlebury, Connecticut
  - 511.74.01009 Boehringer Ingelheim Investigational Site, West Hartford, Connecticut
  - 511.74.01035 Boehringer Ingelheim Investigational Site, Newark, Delaware
  - 511.74.01039 Boehringer Ingelheim Investigational Site, Coral Gables, Florida
  - 511.74.01019 Boehringer Ingelheim Investigational Site, Gainesville, Florida
  - 511.74.01044 Boehringer Ingelheim Investigational Site, Hollywood, Florida
  - 511.74.01001 Boehringer Ingelheim Investigational Site, Hudson, Florida
  - 511.74.01043 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 511.74.01032 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 511.74.01036 Boehringer Ingelheim Investigational Site, Roswell, Georgia
  - 511.74.01047 Boehringer Ingelheim Investigational Site, Champaign, Illinois
  - 511.74.01038 Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - 511.74.01014 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 511.74.01007 Boehringer Ingelheim Investigational Site, Baton Rouge, Louisiana
  - 511.74.01024 Boehringer Ingelheim Investigational Site, Rockland, Maine
  - 511.74.01030 Boehringer Ingelheim Investigational Site, Ann Arbor, Michigan
  - 511.74.01056 Boehringer Ingelheim Investigational Site, Bingham Farms, Michigan
  - 511.74.01010 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 511.74.01012 Boehringer Ingelheim Investigational Site, Billings, Montana
  - 511.74.01045 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 511.74.01041 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 511.74.01055 Boehringer Ingelheim Investigational Site, Reno, Nevada
  - 511.74.01018 Boehringer Ingelheim Investigational Site, Poughkeepsie, New York
  - 511.74.01011 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 511.74.01048 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 511.74.01021 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 511.74.01042 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 511.74.01050 Boehringer Ingelheim Investigational Site, Edmond, Oklahoma
  - 511.74.01006 Boehringer Ingelheim Investigational Site, Eugene, Oregon
  - 511.74.01034 Boehringer Ingelheim Investigational Site, Medford, Oregon
  - 511.74.01040 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 511.74.01017 Boehringer Ingelheim Investigational Site, Anderson, South Carolina
  - 511.74.01057 Boehringer Ingelheim Investigational Site, Knoxville, Tennessee
  - 511.74.01008 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 511.74.01016 Boehringer Ingelheim Investigational Site, Plano, Texas
  - 511.74.01020 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 511.74.01005 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 511.74.01026 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 511.74.01037 Boehringer Ingelheim Investigational Site, Renton, Washington
  - 511.74.01028 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 511.74.01049 Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin
- Canada (10):
  - 511.74.02011 Boehringer Ingelheim Investigational Site, Coquitlam, British Columbia
  - 511.74.02009 Boehringer Ingelheim Investigational Site, Kelowna, British Columbia
  - 511.74.02012 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 511.74.02006 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 511.74.02004 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 511.74.02010 Boehringer Ingelheim Investigational Site, Kingston, Ontario
  - 511.74.02003 Boehringer Ingelheim Investigational Site, Oakville, Ontario
  - 511.74.02002 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 511.74.02007 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 511.74.02008 Boehringer Ingelheim Investigational Site, Montreal, Quebec